CLINICAL TRIAL: NCT00469625
Title: A Study Of Oral Paricalcitol To Treat Proteinuric Renal Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left the Institution.
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Steven Fishbane, MD, Winthrop-University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Z # 13178
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Proteinuric Renal Disease
MeSH Terms: interventions — paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: paricalcitol (initial dose 1 mcg orally per day)

SUMMARY:
Diabetic Nephropathy and other proteinuric renal diseases are the major cause of kidney disease in the United States. The degree of proteinuria is associated with risk for renal disease progression and cardiovascular outcomes. Deficiency of 1-25 Vitamin D develops early in CKD, and is undertreated. Vitamin D may have important effects on factors that drive proteinuria and renal disease progression in patients with proteinuric renal diseases. Therefore, Paricalcitol treatment may reduce proteinuria and slow renal deterioration.

DETAILED DESCRIPTION:
Objectives:

1. To determine the effect of oral paricalcitol on protein excretion in patients with proteinuric renal diseases
2. To determine the effect of oral paricalcitol on renal disease progression in patients with proteinuric renal diseases Hypothesis: Oral paricalcitol will reduce protein excretion in proteinuric kidney disease Study Design: Prospective, randomized, placebo controlled, double blind, trial of paricalcitol compared to placebo.

Sample Size: 60 patients, 30 in each group Summary of Patient Eligibility Criteria: Subjects with proteinuric renal disease (>400 mg/24 hours)

Randomization and Dosage: Patients will be randomized to treatment with oral paricalcitol (initial dose 1 mcg orally per day) compared to placebo Duration : 6 Months

ELIGIBILITY:
Inclusion Criteria:

1. Stable chronic kidney disease
2. Urine protein : Creatinine ratio > 0.4
3. Chronic kidney disease stage 2-4 with eGFR 15-90 ml/min
4. PTH (intact) >20 pg/ml and <250 pg/ml
5. Age 18-85
6. If on ACEI/ARB, then dose optimized (BP, K)

Exclusion Criteria:

1. Failure to provide informed consent
2. Glomerunephritis requiring active treatment with immunosuppresive therapy
3. Serum phosphorus > 5.2
4. Serum calcium (adjusted for albumin)> 10.0
5. Active malignancy
6. Likelihood of requiring renal replacement therapy within 1 year
7. Uncontrolled hypertension

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Winthrop Univ. Hospital, Mineola, New York, United States

REFERENCES:
- [Derived] Fishbane S, Chittineni H, Packman M, Dutka P, Ali N, Durie N. Oral paricalcitol in the treatment of patients with CKD and proteinuria: a randomized trial. Am J Kidney Dis. 2009 Oct;54(4):647-52. doi: 10.1053/j.ajkd.2009.04.036. Epub 2009 Jul 12. PMID 19596163